CLINICAL TRIAL: NCT00666081
Title: A Phase I Open-label Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Potential Anti-cancer Activity of the AKT Inhibitor GSK690693 in Subjects With Relapsed or Refractory Hematologic Malignancies
Brief Title: Study to Investigate AKT Inhibitor GSK690693 in Subjects With Relapsed or Refractory Hematologic Malignancies
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study Cancelled before enrollment
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AKT108169
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Cancer
Keywords: Pazopanib, paclitaxel, carboplatin
MeSH Terms: conditions — Neoplasms | interventions — GSK690693

ARMS (1):
- Cohort 1 (Experimental): GSK690693 for injection. This is a dose escalation study.
  Interventions: Drug: GSK690693

INTERVENTIONS:
Drug: GSK690693 — Administered intravenously at a concentration between 0.1 - 4.8 mg/mL by slow infusion over 4 h.

SUMMARY:
This is a two-part study in subjects with hematologic malignancies designed to find the maximum tolerated dose (MTD) of GSK690693 (Part 1). Part 2 is designed to determine the efficacy of GSK690693 in a subset of subjects with hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically-confirmed diagnosis of a hematologic malignancy that has relapsed or is refractory after standard therapy, AND that is not associated with human immunodeficiency virus (HIV) infection or solid organ transplant.
* Signed written consent provided.
* At least 18 years of age.
* A woman is eligible to enter and participate in the study if she is of: Non-childbearing potential , or is post-menopausal .
* A man with a female partner of childbearing potential is eligible to enter and participate in the study if he has either had a prior vasectomy or agrees to use adequate contraception (as described above) during the study, and up to 3 months after last dose of study drug.
* Fasting glucose that is not elevated.
* Laboratory values within ranges defined in the protocol

Exclusion Criteria:

* Previously diagnosed diabetes mellitus (type 1 or 2), or gestational diabetes.
* Symptomatic or untreated central nervous system (CNS) involvement by the hematologic malignancy (including primary CNS lymphoma). Subjects who were previously treated for CNS involvement, and are asymptomatic without anti-epileptic medications or steroids for at least 2 months are eligible.
* Subjects who have undergone an allogeneic stem cell transplant.
* Unresolved toxicity from previous anti-cancer therapy as agreed to by Medical Monitor and the Investigator,.
* Major surgery within the past 28 days.
* Chemotherapy, radiotherapy, immunotherapy, or investigational drug therapy within 21 days (or 42 days for prior nitrosoureas or mitomycin C) prior to the first dose of study medication. For subjects with acute leukemia, anti-cancer chemotherapy (including corticosteroids) may be administered up to 7 days prior to the first dose of study medication. Chemotherapy given at a dose and schedule that is not expected to have delayed toxicity can be given with an interval of 14 days or more from the first dose. Hydroxyurea may be administered up to 7 days prior to the first dose of study medication.
* Current use of oral corticosteroids, with the exception of inhaled or topical corticosteroids.
* Evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, hepatic, or renal disease).
* Any female who is pregnant or lactating.
* Any serious or unstable pre-existing medical, psychiatric, or other condition (including lab abnormalities) that could interfere with subject safety or with obtaining informed consent.
* Significant ECG abnormalities.
* Use of medications known to prolong the QTc interval within 14 days (or 5 half-lives) prior to the first dose of study medication.
* History of myocardial infarction, acute coronary syndromes, unstable angina or coronary angioplasty/stenting/bypass grafting within the past 6 months.
* Left ventricular ejection fraction (LVEF) less than 50% by echocardiogram (ECHO) or multiple gated acquisition (MUGA) scanning.
* Use of theophylline within 14 days of the first dose of study medication.
* Current use of warfarin ≥4 mg per day; however, low molecular weight heparin and prophylactic low-dose warfarin are permitted, if PT/PTT < 1.2 x ULN.
* Concurrent condition that in the Investigator's opinion would jeopardize the subject's ability to comply with the protocol.
* History of allergic reactions attributed to compounds of similar chemical composition to GSK690693.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
To characterize a range of doses and to identify the MTD of GSK690693 when dosed daily for 5 consecutive days every 21 days as an IV infusion over 4 h. | 21 days

SECONDARY OUTCOMES:
Plasma pharmacokinetic parameters of GSK690693. To evaluate the response of refractory hematologic malignancies to treatment with GSK690693. | 21 days
Blood levels of GSK690693 to derive pharmacokinetic parameters | 21 days
Tumor responses | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline